CLINICAL TRIAL: NCT05624307
Title: Relevance of the Combined Extension-rotation-lateral Tilt Maneuver in the Selection of Patients With Chronic Low Back Pain for Neurotnomy Intervention Radiofrequency : Pilot Study
Brief Title: Selection of Chronic Low Back Pain Patients for Neurotomy Surgery Radiofrequency
Acronym: RaFr
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: FondationbHopale (Other)
Responsible Party: Sponsor
Other Study IDs: HOP22-RIPH3-02
Record Dates: First submitted 2022-11-14; First posted 2022-11-22 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-10

CONDITIONS: Pain;Back Low;Chronic
Keywords: Radiofrequency; Facet pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with chronic back pain: Patients admitted to the chronic pain service at the Calot Institute with chronic low back pain for at least three months, not responding to well-conducted conservative treatment

SUMMARY:
Chronic low back pain is one of the leading causes of disability associated with significant health care costs. One possible management of chronic low back pain of facet origin is neurotomy-radiofrequency (NT-RF) intervention. Currently, to determine whether a patient is eligible for NT-RF, two positive block tests are required.

Clinical examination with a homolateral extension-rotation-tilt maneuver of the spine (ERI maneuver) would have the potential to identify subjects with pain of facet origin. It could therefore be a simple and effective diagnostic tool in the evaluation of a patient with low back pain and help in the decision whether or not to perform a test block by local infiltration of the zygapophyseal joint prior to an NT-RF procedure.

The purpose of this longitudinal, prospective, observational, single-center study is to evaluate the performance of the combined extension-rotation-lateral tilt maneuver (ERI maneuver) in predicting the response to neurotomy-radiofrequency intervention in patients with chronic low back pain.

The included patients will answer 5 questionnaires, in addition to the usual clinical data:

* Hospital Anxiety and Depression scale (HAD) questionnaire,
* Quality of life questionnaire EQ-5D-5L,
* Brief Pain Inventory - French version: Questionnaire Concis de la Douleur (QCD),
* Functional Impotence Scale for Low Back Pain: The Quebec Back Pain Disability Scale
* Clinical Global Impression of Change (CGI-C)

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the chronic pain service at the Calot Institute with chronic low back pain for at least three months, not responding to well-conducted conservative treatment
* Age 18 - 65 years
* Patient did not object to the use of their data
* Patient affiliated to a social security plan

Non inclusion Criteria:

* Patient with a disorder of hemostasis
* Patient with a history of arthrodesis
* Patient with radiologically visible root damage
* Patient with instability of the spine
* Patient with an abnormality on dorso-lumbar MRI: MODIC 1
* Patient under legal protection :

  * Person under guardianship,
  * Person under curatorship,
  * Person under legal protection,
  * Person deprived of liberty,
* Pregnant or breastfeeding woman

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients included in the study were major patients with chronic low back pain.
  The patients included in the study will have to respond to 5 questionnaires at 1 month, 3 months and 6 months according to the frequency of post-treatment consultation with RT-NF.
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2023-11-15 (Estimated); Study Completion 2024-05-15 (Estimated)

PRIMARY OUTCOMES:
Brief-Pain Inventory (BPI) | Pre-operative evaluation, at 1 month
  Patients will be considered responders if the pain score, estimated by the Brief-Pain Inventory (BPI), is reduced by 50% at 1 month compared to the preoperative workup, and non-responders if the pain score did not reduce sufficiently or if the response to block tests was negative.
  Each item is rated from 0, no pain, to 10, pain as bad as you can imagine, and contributes with the same weight to the final score, ranging from 0 to 40. The seven sub-items are rated from 0, does not interfere, to 10, completely interferes, and contributes with the same weight to the final score, ranging from 0 to 70.

SECONDARY OUTCOMES:
The Quebec Back Pain Disability Scale. | Pre-operative evaluation then at 1, 3 and 6 months post intervention
  It is a self-assessment scale of disability, which deals with the impact on daily life and low back pain. It has 20 items, scored from 0 to 5, giving an overall score. The higher the score, the greater the functional impact of low back pain. This scale is validated in French.
Questionnaire Hospital Anxiety and Depression scale (HAD) | Pre-operative evaluation then at 1, 3 and 6 months post intervention
  The Hospital Anxiety and Depression scale (HAD) questionnaire is used to screen for anxiety and depressive disorders. It includes 14 items rated from 0 to 3. Seven questions relate to anxiety (total A) and seven others to the depressive dimension (total D), thus making it possible to obtain two scores (maximum score for each score: 21). A score close to 0 means no anxiety symptoms a score close to 11 and above indicates anxiety symptoms. This scale is validated in French.
EQ-5D-5L Questionnaire | Pre-operative evaluation then at 1, 3 and 6 months post intervention
  The EQ-5D-5L consists essentially of 2 pages: the EQ-5D descriptive system and the EQ Visual Analog Scale (EQ VAS).
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems.
  The EQ VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled 'The best health you can imagine' scored 100 and 'The worst health you can imagine' scored 0. The VAS can be used as a quantitative measure of health outcome that reflect the patient's own judgement.
Brief-Pain Inventory (BPI) | 3 and 6 months post intervention
  Patients will be considered responders if the pain score, estimated by the Brief-Pain Inventory (BPI). Each item is rated from 0, no pain, to 10, pain as bad as you can imagine, and contributes with the same weight to the final score, ranging from 0 to 40. The seven sub-items are rated from 0, does not interfere, to 10, completely interferes, and contributes with the same weight to the final score, ranging from 0 to 70.
  Evolution of BPI scores at 3 and 6 months in patients who responded to treatment at 1 month

OTHER OUTCOMES:
Clinical Global Impression questionnaire (CGI-C) | Pre-operative evaluation then at 1, 3 and 6 months post intervention
  With the Clinical Global Impression (CGI) scale, the physician assesses on a seven-point scale the improvement in the patient's clinical condition following treatment.
  A score of 1 indicates strong improvement and a score of 7 indicates strong clinical worsening of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas OLIVIERI, Principal Investigator — Hopale Foundation - Calot Institute
Locations (1):
- Bruno VEYS, Berck, Hauts-de-France, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://doi.org/10.1097/00007632-199702150-00015
- See also: Related Info — https://doi.org/10.1097/BRS.0b013e3181a1390d
- See also: Related Info — https://doi.org/10.1097/ALN.0000000000002274
- See also: Related Info — https://doi.org/10.7150/ijms.7.124
- See also: Related Info — https://doi.org/10.1097/01.ajp.0000120792.69705.c9
- See also: Related Info — https://doi.org/10.1097/ALN.0b013e3181e33ae5
- See also: Related Info — https://doi.org/10.1016/j.spinee.2006.01.004
- See also: Related Info — https://doi.org/10.1016/j.nephro.2009.01.007